CLINICAL TRIAL: NCT01088243
Title: Targeting Oxidative Stress in Chronic Beryllium Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Lisa Maier, Associate Professor of Medicine, National Jewish Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-2360B
Record Dates: First submitted 2010-03-15; First posted 2010-03-17 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Chronic Beryllium Disease
Keywords: Berylliosis; Beryllium Disease
MeSH Terms: conditions — Berylliosis | interventions — Mesalamine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesalamine (Experimental): Mesalamine (5-ASA) 500 mg capsules four times per day for 6 weeks in Chronic Beryllium Disease subjects.
  Interventions: Drug: Mesalamine
- Placebo (Placebo Comparator): Sugar pill 500 mg capsules four times per day for 6 weeks in Chronic Beryllium Disease subjects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesalamine — Mesalamine (5-ASA) 500 mg capsules four times per day for 6 weeks in Chronic Beryllium Disease subjects.
  Other Names: Pentasa; 5-ASA
  Arms: Mesalamine
Drug: Placebo — Sugar pill 500 mg capsules four times per day for 6 weeks in Chronic Beryllium Disease subjects.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to understand if a drug called mesalamine helps to control inflammation associated with chronic beryllium disease (CBD). We hypothesize that in CBD subjects treated with prednisone, mesalamine treatment will enhance the immunosuppressive effects of prednisone, and thus reduce the immune response to beryllium.

DETAILED DESCRIPTION:
The overall goal of this study is to understand the role of oxidative stress as a potential therapeutic target in the pathogenesis of chronic beryllium disease (CBD). CBD is an inflammatory hypersensitivity lung disease that occurs in an estimated 800,000 beryllium-exposed workers in the United Sates. CBD is characterized by the presence of pulmonary non-caseating granulomas with accumulation of macrophages and beryllium specific CD4+ T cells (Newman et al. 1998). Upon beryllium stimulation in vitro, beryllium specific CD4+ T cells proliferate and produce Th1 cytokines (i.e. TNF-α, IFN-γ, and IL-2) at unusually high levels (Tinkle et al. 1997). The molecular mechanism(s) by which beryllium regulates the chronic production of these cytokines is unknown. Exciting preliminary studies indicate that beryllium alters the redox status of T cells which may adversely modulate the immune response in CBD. Based on these points, a novel hypothesis is proposed: 1) oxidative stress enhances the T cells response to antigen and this enhancement may explain both the excessive cytokine response and the pathogenesis of pulmonary granulomas in CBD and; 2) an inherent difference in T cell antioxidant status is a critical factor in the pathogenesis of CBD. This proposal is a pilot clinical trial examining an approved drug for the treatment of ulcerative colitis (5-amino salicylic acid, 5-ASA), which has anti-inflammatory and antioxidant properties, as a potential new approach for CBD treatment. In this clinical trial, 40 CBD subjects already treated with prednisone, will be treated with either placebo or 5-ASA to determine it effects on the beryllium stimulated immune response in the lung by undergoing bronchoscopy with bronchoalveolar lavage and in blood by undergoing venipuncture before and after 6 weeks of treatment with 5-ASA. As a secondary outcome, we will also assess subjects clinical response to this short course of 5-ASA using spirometry. Bronchoscopies are optional. Patients have the option to participate by undergoing venipuncture and lung function tests only.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic beryllium disease based on the criteria below:

  1. History of beryllium exposure, and;
  2. Positive blood and/or bronchoalveolar lavage Beryllium Lymphocyte Proliferation Tests (BeLPT), and;
  3. Biopsy-proven pathologic changes consistent with CBD-non-caseating granulomas and/or mononuclear cell interstitial infiltrates, and;
  4. Positive bronchoalveolar lavage (BAL) BeLPT and > 15% lymphocytes in BAL fluid.

Exclusion Criteria:

* History of Hepatic disease
* History of Renal disease
* Hypersensitivity to Pentasa (5-ASA) or salicylates.
* Pregnancy
* Presence of another disease that may be expected to significantly affect patient mortality (e.g., HIV), severe cor pulmonale);
* The use of blood thinners.
* Current use of tobacco (smoking or otherwise) in the past 6 months
* Patient inability to participate in the study, such as inability to undergo venipuncture and BAL procedures (if undergoing bronchoscopy) that form part of the inclusion/exclusion criteria or part of the outcome measure.

If undergoing bronchoscopy:

* Severe room air hypoxemia (precluding transbronchial lung biopsy and/or BAL), e.g., pO2 < 45 (Denver altitude 5,280 feet);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Maier, M.D., MSPH, Principal Investigator — National Jewish Health; Brian Day, PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mesalamine | Placebo
Started | 13 | 5
Completed | 12 | 5
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mesalamine | Placebo | Total
Number analyzed (Participants) | 13 | 5 | 18
Age, Continuous [Mean (Full Range); unit: years] | 63.3 [53 to 74] | 62.8 [49 to 79] | 63.16 [49 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 11 | 4 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 5 | 18
Smoking Status [Number; unit: Count of Participants]
  Never | 5 | 2 | 7
  Former | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Beryllium Lymphocyte Proliferation Responses (BeLPT) From Baseline to Week 6
Description: Primary endpoints are beryllium proliferation responses (BeLPT) in PBMCs (peripheral blood mononuclear cells) and BAL (bronchoalveolar lavage) cells. The BeLPT is a blood test that measures the immune response to beryllium exposure. If immune cells multiply in response to beryllium, this is considered an abnormal test results. If immune cells do not multiple, this is considered a normal test results. Results are reported as "stimulation index", which is a ratio of the number of cells grown with beryllium compared to the number of cells grown without beryllium. A value of 2.5 or less is considered normal, and a value greater than 2.5 is abnormal.
Time Frame: baseline and week 6
Population: Because bronchoscopy was not required for participation, only three placebo and six 5-ASA-treated subjects underwent bronchoscopy and is reported under BAL.
Measure: Mean (Standard Deviation); unit: Stimulation index
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 13 | 5
Stimulation index
  BAL: number analyzed (Participants) | 6 | 3
  BAL | 48.61 (57.18) | 9.33 (14.08)
  PBMC | 22.07 (20.30) | 3.8 (6.09)

2. Secondary Outcome: Changes in Bronchoalveolar Lavage (BAL) Tumor Necrosis Factor Alpha (TNFa)
Description: Secondary outcomes include changes in bronchoalveolar lavage (BAL) tumor necrosis factor alpha (TNFa)
Time Frame: baseline and week 6
Population: We did not have sufficient cells to run experiments on all participants. However, below is a summary of what data was received.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 6 | 3
pg/ml | 62 (35.76) | -1750 (2734)

3. Secondary Outcome: Changes in Steady-state Glutathione (GSH) Levels From Baseline to Week 6
Description: Secondary outcomes include changes in steady-state GSH levels in beryllium specific CD4+ T cell in bronchoalveolar lavage fluid (BALF)
Time Frame: baseline and week 6
Population: We did not receive enough cells from participants to be able to run experiments on all. However, below is a summary of what data was received.
Measure: Mean (Standard Deviation); unit: mmol/mg
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 6 | 3
mmol/mg | 4.93 (20.08) | 10.38 (16.5)

4. Secondary Outcome: HDAC2 Levels
Description: Secondary outcomes include changes in HDAC2 levels
Time Frame: baseline and week 6
Population: We were not able to perform due to insufficient samples and data collected from each participant to summarize changes in HDAC2 levels.
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Glucocorticoid Receptors
Description: Secondary outcomes include changes in glucocorticoid receptors modification in PBMCs and BAL cells.
Time Frame: baseline and week 6
Population: We were not able to perform due to insufficient samples and data collected from each participant to summarize changes.
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Lung Function
Description: Secondary outcomes include changes in lung function, which will be assessed with Forced expiratory volume in 1 second percent predicted (FEV1), Forced vital capacity percent predicted (FVC) and Diffusing capacity percent predicted (DLCO).
Time Frame: baseline and week 6
Population: One participant did not complete follow up in Mesalamine group. However, below is a summary of what data was received.
Measure: Mean (Standard Deviation); unit: percentage of predicted value
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 12 | 5
percentage of predicted value
  FEV1 % pred | 2.2 (4.49) | -0.91 (4.73)
  FVC % pred | 1.6 (3.5) | -0.08 (5.55)
  DLCO % pred | 2.4 (4.39) | -0.16 (6.01)

ADVERSE EVENTS:
Time Frame: The patients will be monitored after baseline evaluation, during drug therapy, and after 2 week follow-up evaluation by a study coordinator and Dr. Maier who will follow-up for adverse events at each visit. All adverse events (serious and moderate/mild) associated with bronchoscopy procedures and study drug will be assessed individually by study PIs for appropriate action if necessary.
Arm/Group | Mesalamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/5
Other Adverse Events (participants affected / at risk) | 2/13 | 2/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesalamine (N=13) | Placebo (N=5)
Mobitz Type II heart block (Cardiac disorders) | 0 (0) | 1 (1) — In the placebo-treated subjects, we identified a Mobitz Type II heart block during a follow-up bronchoscopy. It was not related to the treatment.
Swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
One 5-ASA-treated subject developed dizziness, constipation, stomach pain and chest pain two weeks (General disorders) | 1 (1) | 0 (0) — Dizziness, constipation, stomach pain and chest pain
One 5-ASA-treated subject experienced coughing and low energy after the follow-up bronchoscopy (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No